CLINICAL TRIAL: NCT01706159
Title: A Multicenter, Randomised, Double-blind, Placebo-controlled, Multiple-dose Trial With rFXIII Administered to Subjects With Mild to Moderate Active Ulcerative Colitis
Brief Title: A Placebo-controlled Trial With rFXIII Administered to Subjects With Mild to Moderate Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial screening data did not support the medical hypothesis
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8717-3946; 2011-001568-22 (EudraCT Number); U1111-1120-3824 (Other: WHO)
Record Dates: First submitted 2012-10-09; First posted 2012-10-15 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Inflammation; Ulcerative Colitis
MeSH Terms: conditions — Inflammation; Colitis, Ulcerative | interventions — recombinant factor XIII-A2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog
- Placebo (Active Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — Catridecacog (recombinant factor XIII, rFXIII) will be administered as intravenous (i.v.) injections (at an approximate rate of 1-2 mL/min) once every second week at a dose of 35 IU/kg
  Other Names: recombinant factor XIII
  Arms: rFXIII
Drug: placebo — Placebo will be administered as intravenous (i.v.) injections (at an approximate rate of 1-2 mL/min) once every second week.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the effect of recombinant factor XIII (rFXIII) administered to subjects with mild to moderate active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ulcerative colitis for at least 3 months from the time of initial diagnosis. The diagnosis must have been confirmed by historical endoscopy and histology. The severity of disease must have been confirmed by endoscopy at screening
* Currently receiving oral aminosalicylates at approved doses of at least 2g/day for at least 6 weeks. Doses of oral aminosalicylates should be stable for at least two weeks prior to dosing (Visit 2)

Exclusion Criteria:

* Diagnosis of UC limited to the rectum (ulcerative proctitis only, defined as less than 15 cm from the anal verge)
* Requiring hospitalisation for current episode of severe UC
* Use of biologic therapies for the treatment of UC within 12 weeks prior to dosing (Visit 2)
* Treatment failures to anti-tumour necrosis factor-alfa (anti-TNF-a) agents (e.g. infliximab, adalimumab)
* Use of immunosuppressant agents (e.g. azathioprine) within 4 weeks prior to dosing (Visit 2)
* Use of corticosteroids (oral, intravenous (i.v.), intramuscular (i.m.), or rectal ) within 14 days prior to dosing (Visit 2)
* Use of enemas (corticosteroid or aminosalicylate) within 14 days prior to screening (Visit 1)
* Use of cyclosporine, tacrolimus, D-penicillamine, leflunomide, methotrexate, mycophenolate mofetil, or thalidomide within 4 weeks prior to dosing (Visit 2)
* Currently receiving total parenteral nutrition

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- Rousse, Bulgaria
- Zagreb, Croatia
- Herlev, Denmark
- Békéscsaba, Hungary
- Lodz, Poland
- Nizhny Novgorod, Russia
- Kharkiv, Ukraine

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 12 sites in 6 countries as follows: Bulgaria (4 sites), Denmark (1 site), Hungary (1 site), Poland (4 sites), Russian Federation (1 site) and Ukraine (1 site).
Pre-assignment Details: No pre-assignments were given for this trial.
Groups:
- rFXIII: Recombinant factor XIII (rFXIII) was administered as intravenous (i.v.) injections (at an approximate rate of 1-2 mL/min) at a dose of 35 IU/kg. The doses were administered once every second week for a total of 4 doses.
- Placebo: Placebo formulation was administered as intravenous (i.v.) injections (at an approximate rate of 1-2 mL/min) once every second week. The doses were administered for a total of 4 doses.
Period: Overall Study
Arm/Group | rFXIII | Placebo
Started | 14 | 6
Exposed | 13 (One subject was not exposed to rFXIII.) | 5 (One subject was not exposed to placebo.)
Completers (With Baron Score at Week 8) | 6 | 3
Completed | 6 | 4
Not Completed | 8 | 2
Not completed — Withdrawal Criteria | 2 | 1
Not completed — Unclassified | 6 | 1

BASELINE CHARACTERISTICS:
Population: The demographics and baseline characteristics are presented for the Full analysis set (FAS) which included all randomised and treated subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | rFXIII | Placebo | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (10.6) | 45.0 (15.4) | 39.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 1 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Whites | 13 | 5 | 18
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.5 (3.2) | 25.6 (5.8) | 24.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Remission Defined as a Modified Baron Score of 0
Description: The primary endpoint was the binary variable ("responder" vs. "non-responder") where "responders" were the subjects with endoscopic remission (endoscopic mucosal healing) at Week 8, defined as a modified Baron score of 0. Subjects with a modified Baron score ≥1 were designated as "non-responders".
Time Frame: At week 8
Population: Full analysis set (FAS) included all randomised and treated subjects.
Measure: Number; unit: Subjects
Arm/Group | rFXIII | Placebo
Number analyzed (Participants) | 13 | 5
Subjects | 1 | 1
Statistical Analysis 1: Comparison: rFXIII vs Placebo; A sample size of 90 subjects, with a 2:1 (active:placebo) randomization ratio, would ensure 80% power to detect a difference between active treatment and placebo at Week 8 with a 2-sided significance level of 10% based on a Fisher's exact test; Test type: Superiority or Other; p = 0.3056, Regression, Logistic — p-value was not adjusted for multiple comparisons; Odds Ratio (OR) = 0.16, 90% CI [0.01 to 3.05]

2. Secondary Outcome: Remission (Clinical and Endoscopic)
Description: Analysis of responders defined by a clinical component of: ulcerative colitis disease activity index (UC-DAI) score of less than or equal to 1 with 0 for rectal bleeding and 0 for stool frequency and an endoscopic component of: no mucosal friability (modified Baron score less than or equal to 1).
Time Frame: At Week 8
Population: Full analysis set (FAS) included all randomised and treated subjects. Two subjects in the rFXIII group had no UC-DAI score at any visit, including baseline and they were excluded from the analysis.
Measure: Number; unit: Subjects
Arm/Group | rFXIII | Placebo
Number analyzed (Participants) | 11 | 5
Subjects | 0 | 0

3. Secondary Outcome: Number of Adverse Events (AEs)
Description: Number of adverse events reported from the first trial-related activity, after the subject was exposed to the trial drug, until the end of the post-treatment follow-up period.
Time Frame: Week 0 to 10
Population: Safety analysis set included all randomised and treated subjects.
Measure: Number; unit: events
Arm/Group | rFXIII | Placebo
Number analyzed (Participants) | 13 | 5
events
  Adverse events | 7 | 4
  Serious adverse events | 1 | 0
  Severe adverse events | 1 | 0
  Moderate adverse events | 0 | 2
  Mild adverse events | 6 | 2
  Fatal adverse events | 0 | 0

4. Secondary Outcome: Clearance (CL) of rFXIII
Description: The volume of plasma cleared of the drug per unit time.
Time Frame: Samples were collected before and up to 72 hours after the first dose of rFXIII.
Population: It was not possible to obtain credible single dose pharmakokinetics (PK) for rFXIII in this trial due to a small number of subjects with required PK measurements and a spurious behaviour of individual PK profiles.
Arm/Group | rFXIII | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Maximum Concentration (Cmax) of rFXIII
Description: The peak plasma concentration of the drug after dose administration.
Time Frame: Samples were collected before and up to 72 hours after the first dose of rFXIII.
Population: It was not possible to obtain credible single dose PK for rFXIII in this trial due to a small number of subjects with required PK measurements and a spurious behaviour of individual PK profiles.
Arm/Group | rFXIII | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events reported by the investigator from the first trial-related activity after the subject is exposed to the trial drug until the end of trial visit (Week 10).
Description: Safety analysis set was identical to the FAS which included all randomised and treated subjects.
Arm/Group | rFXIII | Placebo
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/5
Other Adverse Events (participants affected / at risk) | 2/13 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII (N=13) | Placebo (N=5)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rFXIII (N=13) | Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated earlier than planned as the hypothesis of a correlation between low levels of FXIII and disease activity of UC could not be confirmed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Novo Nordisk reserves the right to prior review of such publications and to ask for delay of publication of individual site results until after the primary manuscript is accepted for publication.